CLINICAL TRIAL: NCT02811081
Title: The Effective Maneuver to Reduce Shoulder Pain After Laparoscopic Gynecologic Surgery: Randomized Controlled Trial
Brief Title: Effective Maneuver for Post-laparoscopic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoungho Ryu, Clinical assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-05-048
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Gynecologic Diseases
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Passive deflation of residual carbon dioxide
  Interventions: Procedure: Passive Deflation
- Normal Saline Instillation (Experimental): Instillation of isotonic normal saline in the sub-diaphragmatic region
  Interventions: Procedure: Normal Saline Instillation
- Combined Intervention (Experimental): Normal Saline Instillation + Pulmonary Recruitment
  Interventions: Procedure: Normal Saline Instillation + Pulmonary Recruitment

INTERVENTIONS:
Procedure: Passive Deflation — In the control group, residual carbon dioxide gas was evacuated by the routine method using passive exsufflation through the port site at the end of surgery.
  Arms: Control
Procedure: Normal Saline Instillation — In the normal saline instillation group, in addition to the routine method, the patients were placed in the Trendelenburg position (30°), isotonic normal saline (20 ml/kg of body weight) was infused in the sub-diaphragmatic region at the end of surgery.
  Arms: Normal Saline Instillation
Procedure: Normal Saline Instillation + Pulmonary Recruitment — In the combined intervention group, in addition to the routine method, the patients were placed in the Trendelenburg position (30°), and a pulmonary recruitment maneuver was performed after instillation of isotonic normal saline (20 ml/kg of body weight) in the sub-diaphragmatic region at the end of surgery.
  Arms: Combined Intervention

SUMMARY:
The aim of this clinical trial is to estimate the efficacy and safety of combined intervention with the intra-peritoneal normal saline instillation and pulmonary recruitment maneuver for reducing post-laparoscopic shoulder pain.

DETAILED DESCRIPTION:
Shoulder pain after laparoscopy is common and its probable mechanism is residual carbon dioxide gas after surgery. Both the intra-peritoneal normal saline instillation and pulmonary recruitment maneuver could effectively reduce post-laparoscopic shoulder pain. However, the efficacy and safety of combined intervention with normal saline instillation and pulmonary recruitment maneuver have not been investigated yet. The aim of this clinical trial is to estimate the effectiveness of combined intervention with the intra-peritoneal normal saline instillation and pulmonary recruitment maneuver for reducing post-laparoscopic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopy for benign gynecologic diseases
* patients aged 19-65 years
* patients with american society of anesthesiology physical status I-II
* patients obtaining written informed consent

Exclusion Criteria:

* patients with chronic shoulder pain, chronic epigastric pain or chronic pain syndrome
* patients with past history of pneumothorax or any pulmonary surgical history
* patients with any shoulder surgery histories
* patients who required to conversion to open surgery from laparoscopic surgery
* patients who required to receive incidental upper abdominal surgeries due to adhesion and injury at upper abdominal cavity
* patients with inability to understand or express 10 point visual analogue scale
* pregnant women

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Shoulder pain evaluated by 10 point visual analogue scale | after two day of procedure
  The pain score was evaluated by 10 point visual analogue scale.

SECONDARY OUTCOMES:
Wound pain evaluated by 10 point visual analogue scale | after two day of procedure
  The pain score was evaluated by 10 point visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided